CLINICAL TRIAL: NCT03372551
Title: Comparison of Daily Disposable Invigor I (Test) and Select 1 Day Lenses
Brief Title: Comparison of Somofilcon A Daily Disposable Test Contact Lens and Somofilcon A Daily Disposable Control Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CV-16-43
Record Dates: First submitted 2017-12-08; First posted 2017-12-13 (Actual); Results first posted 2019-05-29 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Intervention Model Description: This will be a, prospective, double-masked, randomized, bilateral, 1 week cross-over, dispensing study
Who Masked: Participant, Investigator
Masking Description: Both the participants and study investigators will be masked to the randomization schedule of the contact lenses used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- somofilcon A 1 day test lens (Experimental): Subjects wearing the somofilcon A 1 day test lens for one week, either randomized as the first or second pair.
  Interventions: Device: somofilcon A 1 day test lens; Device: somofilcon A 1 day control lens
- somofilcon A 1 day control lens (Active Comparator): Subjects wearing the somofilcon A 1 day control lens for one week, either randomized as the first or second pair.
  Interventions: Device: somofilcon A 1 day test lens; Device: somofilcon A 1 day control lens

INTERVENTIONS:
Device: somofilcon A 1 day test lens — Contact lens
  Other Names: somofilcon A daily disposable test soft contact lens; Invigor I; Test lens
Device: somofilcon A 1 day control lens — Contact lens
  Other Names: somofilcon A daily disposable control soft contact lens; Select 1-Day; Control lens

SUMMARY:
The purpose of this study is to investigate the overall clinical performance of the somofilcon A daily disposable test soft contact lens compared to the somofilcon A daily disposable control soft contact lens.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the clinical performance of an investigational silicone-hydrogel contact lens (test) against a marketed silicone-hydrogel contact lens (control) when worn on a daily disposable wear modality over 1 week (for each lens) in a randomized, bilateral, cross-over, dispensing study.

ELIGIBILITY:
Inclusion Criteria:

* Is at least 17 years of age and has full legal capacity to volunteer;
* Has had a self-reported oculo-visual examination in the last two years;
* Has read, understood, and signed the information consent letter;
* Is willing and able to follow instructions and maintain the appointment schedule;
* Has a visual acuity of 20/30 or better (in each eye) with their habitual vision correction, or 20/20 best-corrected vision (for binocular distance acuity);
* Must be able to achieve 20/30 or better (in each eye) with the study lenses;
* Currently wears soft contact lenses for at least 3 days per week, 8 hours each day;
* Requires spectacle lens powers between -0.75 and -06.50 diopters sphere (0.25D steps);
* Has no more than 0.75 diopters of refractive astigmatism;
* Has clear corneas and no active* ocular disease;
* Has not worn lenses for at least 12 hours before the examination.

Exclusion Criteria:

* Is presently participating in any other clinical or research study including eye related clinical or research study;
* Has never worn contact lenses before.
* Has any systemic disease affecting ocular health.
* Has any active* ocular pathology or severe insufficiency of lacrimal secretion (moderate to severe dry eyes) that would affect the wearing of contact lenses.
* Is using any systemic or topical medications that will affect a study outcome variable, and/or ocular health.
* Has any known sensitivity to fluorescein dye or products to be used in the study.
* Has persistent, clinically significant corneal or conjunctival staining using sodium fluorescein dye.
* Has any clinically significant lid or conjunctival abnormalities, active neovascularization or any central corneal scars.
* Is aphakic.
* Has undergone corneal refractive surgery.
* Is pregnant, lactating, or planning a pregnancy at the time of enrolment (by verbal confirmation at the screening visit).

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2017-12-22 (Actual); Study Completion 2018-04-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Contact Lens Research, University of Waterloo, Waterloo, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three (3) subjects did not meet inclusion criteria and were excluded from the analysis. One subject was enrolled and later discontinued.
Groups:
- Somofilcon A 1 Day Test Lens First, Then Control 1 Day Lens: Subjects wear the somofilcon A 1 day Test Lens first for one week, then somofilcon A 1 day Control lens for one week.
  somofilcon A 1 day test lens: Contact lens
  somofilcon A 1 day control lens: Contact lens
- Somofilcon A 1 Day Control Lens First, Then 1 Day Test Lens: Subjects wear the somofilcon A 1 day Control lens first for one week, then somofilcon A 1 day Test lens for one week.
  somofilcon A 1 day test lens: Contact lens
  somofilcon A 1 day control lens: Contact lens
Period: First Intervention (1 Week)
Arm/Group | Somofilcon A 1 Day Test Lens First, Then Control 1 Day Lens | Somofilcon A 1 Day Control Lens First, Then 1 Day Test Lens
Started | 17 | 16
Completed | 16 | 16
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Second Intervention (1 Week)
Arm/Group | Somofilcon A 1 Day Test Lens First, Then Control 1 Day Lens | Somofilcon A 1 Day Control Lens First, Then 1 Day Test Lens
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Somofilcon A 1 Day Test vs Control Contact Lens: Each subjects randomized to wear either the test or control as a matched pair and cross over to second matched pair.
  somofilcon A 1 day test lens: Test / Contact lens
  somofilcon A 1 day control lens: Test / Contact lens
Arm/Group | Somofilcon A 1 Day Test vs Control Contact Lens
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 31
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 32
Region of Enrollment [Number; unit: participants]
  Canada | 32

OUTCOME MEASURES:

1. Primary Outcome: Comfort
Description: Subjective comfort scored 0-100 (0=Cannot be worn, 100=Cannot be felt ever)
Time Frame: up to 1 week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Somofilcon A 1 Day Test Lens | Somofilcon A 1 Day Control Lens
Number analyzed (Participants) | 32 | 32
score on a scale
  Comfort at Dispense | 90 (8) | 89 (11)
  Comfort at Insertion after 1 week | 86 (11) | 87 (16)
  Comfort during day after 1 week | 84 (11) | 86 (11)
  Comfort end day after 1 week | 75 (15) | 78 (16)
  Overall comfort after 1 week of lens wear | 82 (11) | 85 (12)

2. Primary Outcome: Preference
Description: Overall lens that subject prefers or no preference
Time Frame: up to 1 week
Measure: Count of Participants; unit: Participants
Groups:
- Somofilcon A 1 Day Test / Control Contact Lens: Each subjects randomized to wear either the somofilcon A 1 day test or somofilcon A 1 day control as a matched pair and cross over to second matched pair.
  somofilcon A 1 day test lens: Test / Contact lens
  somofilcon A 1 day control lens: Test / Contact lens
Arm/Group | Somofilcon A 1 Day Test / Control Contact Lens
Number analyzed (Participants) | 32
Participants
  Strongly preferred somofilcon A 1 Day Test lens | 5
  Slightly preferred somofilcon A 1 Day Test lens | 9
  No preference | 1
  Slightly preferred somofilcon A 1 Day Control lens | 5
  Strongly preferred somofilcon A 1 Day control lens | 12

3. Primary Outcome: Vision
Description: Visual acuity measured in logMAR
Time Frame: Up to 1 week
Population: Dispensing - n=32 participants total, 1 week = 31 participants total due to a nonserious adverse events for somofilcon A 1 day test lens.
Measure: Mean (Standard Deviation); unit: Log(MAR)
Groups:
- Somofilcon A 1 Day Test Lens Dispense; Somofilcon A 1 Day Test Lens 1 Week: Subjects wearing the somofilcon A 1 day test lens for one week, either randomized as the first or second pair.
  somofilcon A 1 day test lens: Contact lens
  somofilcon A 1 day control lens: Contact lens
- Somofilcon A 1 Day Control Lens Dispense; Somofilcon A 1 Day Control Lens 1 Week: Subjects wearing the somofilcon A 1 day control lens for one week, either randomized as the first or second pair.
  somofilcon A 1 day test lens: Contact lens
  somofilcon A 1 day control lens: Contact lens
Arm/Group | Somofilcon A 1 Day Test Lens Dispense | Somofilcon A 1 Day Test Lens 1 Week | Somofilcon A 1 Day Control Lens Dispense | Somofilcon A 1 Day Control Lens 1 Week
Number analyzed (Participants) | 32 | 31 | 32 | 31
Log(MAR)
  High Illumination high contrast monocular | -0.10 (0.07) | -0.10 (0.07) | -0.11 (0.07) | -0.11 (0.06)
  High Illumination high contrast binocular | -0.15 (0.06) | -0.15 (0.07) | -0.15 (0.06) | -0.16 (0.06)
  Low Illumination high contrast monocular | -0.08 (0.05) | -0.07 (0.07) | -0.09 (0.07) | -0.10 (0.06)
  Low Illumination high contrast binocular | -0.13 (0.06) | -0.13 (0.07) | -0.13 (0.06) | -0.14 (0.05)

4. Primary Outcome: Subjective Vision
Description: Subjective vision scored 0-100 (0=Extremely poor, 100=Excellent vision all the time)
Time Frame: up to 1 week
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Somofilcon 1 Day Test Lens: Vision Quality/Clarity During Day: Subjects wearing the somofilcon A 1 day test lens for one week, either randomized as the first or second pair.
  somofilcon A 1 day test lens: Contact lens
  somofilcon A 1 day control lens: Contact lens
- Somofilcon A Control Lens: Vision Quality/Clarity During Day: Subjects wearing the somofilcon A 1 day control lens for one week, either randomized as the first or second pair.
  somofilcon A 1 day test lens: Contact lens
  somofilcon A 1 day control lens: Contact lens
Arm/Group | Somofilcon 1 Day Test Lens: Vision Quality/Clarity During Day | Somofilcon A Control Lens: Vision Quality/Clarity During Day
Number analyzed (Participants) | 32 | 32
score on a scale
  Dispense | 92 (9) | 92 (6)
  1 week | 88 (12) | 91 (11)

5. Primary Outcome: Corneal Staining
Description: Amount of staining observed on the cornea scored 0-4 (0=none, 4=severe) in 0.25 steps
Time Frame: up to 1 week
Population: Baseline n=32 participants / 64 eyes, 1 week n = 31 participants / 62 eyes due to non-serious adverse event participant's measurements weren't completed.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Eye
Arm/Group | Somofilcon A 1 Day Test Lens | Somofilcon A 1 Day Control Lens
Number analyzed (Participants) | 32 | 32
Number analyzed (Eye) | 64 | 64
score on a scale
  Baseline | 0.16 (0.25) | 0.16 (0.25)
  1 week: number analyzed (Participants) | 31 | 31
  1 week: number analyzed (Eye) | 62 | 62
  1 week | 0.20 (0.26) | 0.18 (0.42)

6. Primary Outcome: Conjunctival Staining
Description: Amount of staining observed on the conjunctiva scored 0-4 (0=none, 4=severe) in 0.25 steps
Time Frame: up to 1 week
Population: Baseline n=32 participants / 64 eyes, 1 week n= 31 participants / 62 eyes due to non-serious adverse event participant's measurements weren't completed.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | Somofilcon A 1 Day Test Lens | Somofilcon A 1 Day Control Lens
Number analyzed (Participants) | 32 | 32
Number analyzed (Eyes) | 64 | 64
score on a scale
  Baseline | 0.20 (0.25) | 0.20 (0.25)
  1 week: number analyzed (Participants) | 31 | 31
  1 week: number analyzed (Eyes) | 62 | 62
  1 week | 0.72 (0.57) | 0.91 (0.71)

ADVERSE EVENTS:
Time Frame: From dispense to completion of follow up, up to 2 weeks.
Arm/Group | Somofilcon A 1 Day Test Lens | Somofilcon A 1 Day Control Lens
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 0/32 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure restriction on the PI is that the sponsor should be notified of any results communications and has ability to review.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-20): https://cdn.clinicaltrials.gov/large-docs/51/NCT03372551/Prot_SAP_001.pdf